CLINICAL TRIAL: NCT05741970
Title: Interaction Between Hypertension and Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Nurdan Ozmeric, Professor, Gazi University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: GU291208/11
Record Dates: First submitted 2022-11-16; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Hypertension; Periodontitis
Keywords: IL-6; CRP; Periodontitis; Hypertension; Phase I therapy
MeSH Terms: conditions — Hypertension; Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Examiner who recorded the clinical indexes was blinded to the systemical status of the patients and the periodontologists who were responsible for patients periodontal treatment were not blinded because of the anesthesia applied to hypertension patients and the precautions needed to be taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IL-6 and CRP levels of the hypertensive and periodontitis group (Active Comparator): All patients with periodontitis received phase I periodontal therapy including oral hygiene instruction (OHI) and scaling/root planning (SRP) without any antimicrobial therapy. GCF and saliva samples were obtained and clinical measurements were performed at baseline (before treatment (BT) and four weeks (4 weeks 3 days) after the phase I periodontal therapy (AT).
  Interventions: Procedure: Scaling and root planing
- IL-6 and CRP levels of the hypertensive and healthy group (No Intervention): GCF and saliva samples were obtained and clinical measurements were performed at baseline
- IL-6 and CRP levels of the periodontitis and healthy group (Active Comparator): All patients with periodontitis received phase I periodontal therapy including oral hygiene instruction (OHI) and scaling/root planning (SRP) without any antimicrobial therapy. GCF and saliva samples were obtained and clinical measurements were performed at baseline (before treatment (BT) and four weeks (4 weeks 3 days) after the phase I periodontal therapy (AT).
  Interventions: Procedure: Scaling and root planing
- IL-6 and CRP levels of the systemically and periodontally healthy group (No Intervention): GCF and saliva samples were obtained and clinical measurements were performed at baseline

INTERVENTIONS:
Procedure: Scaling and root planing — Each tooth with inflammation symptoms was cleaned with scalers, curettes and ultrasonic devices routinely.
  Arms: IL-6 and CRP levels of the hypertensive and periodontitis group; IL-6 and CRP levels of the periodontitis and healthy group

SUMMARY:
Objective:The possible association between hypertension and periodontitis and the effect of hypertension on periodontal treatment were investigated by evaluating salivary and gingival crevicular fluid (GCF) interleukin (IL)-6 and C reactive protein (CRP) levels. Methods:Forty two healthy individuals without any previously diagnosed systemic disease [10 periodontally healthy (control) and 10 periodontitis (CP)] and subjects with hypertension [13 periodontally healthy (HP) and 9 with periodontitis (CP + HP)] participated in the study. GCF and saliva samples were obtained at baseline and four weeks after Phase I periodontal treatment. Biochemical parameters were analyzed using ELISA. Results:Before the periodontal treatment, significantly higher GCF IL-6 and CRP levels were detected in CP+HP and CP groups compared to HP and control groups (p<0.01). Salivary CRP level in CP+HP group was found to be higher than the control group (p<0.05). Statistically significant gingival and plaque index measurements (p<0.01) might suggest a possible effect of hypertension on periodontal status. Periodontal treatment significantly improved the clinical indices, however biochemical parameters did not change after the treatment. Conclusion:the association of hypertension with periodontitis through local salivary and GCF mediators might be possible in disease process.

DETAILED DESCRIPTION:
Forty-two participants were included in the study. The study groups consisted of 20 healthy individuals without any previously diagnosed systemic disease (10 periodontally healthy and 10 with periodontitis) and 22 patients with hypertension (13 periodontally healthy and 9 with periodontitis). The patient population was randomly selected among the patients who referred to Periodontology Clinic. Hypertensive patients with at least 5 years of follow up were included in the hypertension group. Hypertension patients treated with antihypertensive drugs known to cause gingival overgrowth were excluded from the study.

Other exclusion criteria were diabetes mellitus, high cholesterol levels, CVD and drugs usage other than antihypertensive drugs. A calibrated examiner performed a comprehensive periodontal examination included plaque index (Silness & Loe, 1964) (PI), gingival index (Loe & Silness, 1963) (GI), probing depth (PD), clinical attachment level (CAL) and bleeding on probing (BOP). The measurements were made at six sites per tooth (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual and disto-lingual) using a periodontal probe (Williams periodontal probe, Nordent Manufacturing, Elk Grove Village, IL., USA) To perform the intra-examiner calibration, PD and CAL were measured twice at six sites of each tooth within 24 hours. Intra-examiner agreement was at least 90% for both PD and CAL within 1 mm. Examiner who recorded the clinical indexes was blinded to the systemical status of the patients and the periodontologists who were responsible for patients periodontal treatment were not blinded because of the anesthesia applied to hypertension patients and the precautions needed to be taken.

During the study period, patients were instructed not to use any local/systemic antibiotics and antimicrobial agents.Patients diagnosed with periodontitis had Stage II periodontitis in a generalized pattern with probing depths of 3-4mm. The diagnosis was performed based on criteria that maximum probing depth ≤5 mm, mostly horizontal loss and >30% of teeth involved. Healthy periodontium was identified as the presence of BOP≤10% and PD≤3 mm.The deepest four pockets of non-adjacent single rooted teeth were selected for GCF sampling. The participants were distributed into four groups; healthy subjects with healthy periodontal condition (control), healthy subjects with periodontitis (CP), hypertension patients with periodontitis (CP + HP) and hypertension patients with healthy periodontal condition (HP). The study was approved by the local ethics committee (291208/11) and all patients signed an informed consent form. Exclusion criteria were smoking, pregnancy, established secondary hypertension diagnosis, other systemic diseases and previous periodontal and/or antibiotic treatment within the last six months. All patients with periodontitis received phase I periodontal therapy including oral hygiene instruction (OHI) and scaling/root planning (SRP) without any antimicrobial therapy. GCF and saliva samples were obtained and clinical measurements were performed at baseline (before treatment (BT) and four weeks after the phase I periodontal therapy (AT). The timeline for the phase I therapy (within 2 weeks of baseline examination 4 days). Primary biochemical outcome measures included salivary and GCF IL-6 and CRP, and primary periodontal outcome measures were PI, GI, PD, CAL and BOP. Secondary outcome measure was GCF volume.

GCF and saliva sampling and processing The GCF sampling site was gently air dried and supragingival plaque was removed.

The area was carefully isolated with cotton rolls in order to prevent contamination.

Standardized paper strips (Periopaper, Pro Flow, Amityville, NY, USA) were inserted into the sulcus until slight resistance was felt and left in place for 30 seconds. Strips contaminated by bleeding or exudates were discarded. GCF volumes were determined as described previously. To determine the amount of GCF, an electronic balance was used to weigh the paper strips before and immediately after collection. The mass (mg) of the fluid on each strip was converted to a volume in millimeters by assuming that the density of GCF was 1. Strips were placed into coded micro centrifuge tubes and stored at -800C until processing. Before biochemical analysis, paper strips were placed in 0,1 % bovine serum albumin/phosphate buffered saline solution in Eppendorf tubes, and the fluid from the paper strip was eluted by centrifugation for 6 minutes at 5,000 · g at 4 C. Following centrifugation, the strips were removed.The participants were asked to stop eating and drinking 2 hours before each sampling. They were instructed to rinse their mouth for 30 seconds with 10 mL of water and to rest for 2 minutes before unstimulated saliva was collected by spitting. Approximately 1 mL of unstimulated whole saliva was collected into Eppendorf tubes. Samples were centrifuged for 10 minutes at 15.000 × g at 4°C to remove any particulate matter. The supernatants were stored at -20°C until analysed.

GCF and saliva enzyme-linked immunosorbent assay (ELISA) analysis for IL-6 and CRPThe levels of IL-6 and CRP in GCF and saliva were measured using a sandwich ELISA kit (Biosource, Invitrogen Corporation, Carlsbad, California 92008). The ELISA procedures were carried out according to the manufacturer's instructions. Results were expressed as pg/mL. Total amounts were also calculated by multiplying concentrations and CRP volumes.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients with at least 5 years of followup were included in the hypertension group.

Exclusion Criteria:

* Hypertension patients treated with antihypertensive drugs known to cause gingival overgrowth were excluded from the study.

Other exclusion criteria were diabetes mellitus, high cholesterol levels, CVD and drugs usage other than antihypertensive drugs.

Ages: 39 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Salivary and Gingival crevicular fluid Interleukin-6 and CRP | change from baseline to postoperative 4 weeks
  pg/mL unite
Plaque index and Gingival index | change from baseline to postoperative 4 weeks
  scores from 1-3
Pocket depth and Clinical attachment level | change from baseline to postoperative 4 weeks
  mm
Bleeding on probing | change from baseline to postoperative 4 weeks
  percentage

SECONDARY OUTCOMES:
Gingival crevicular fluid volume | change from baseline to postoperative 4 weeks
  microgram

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bengtsson VW, Persson GR, Berglund JS, Renvert S. Periodontitis related to cardiovascular events and mortality: a long-time longitudinal study. Clin Oral Investig. 2021 Jun;25(6):4085-4095. doi: 10.1007/s00784-020-03739-x. Epub 2021 Jan 28. PMID 33506429
- [Result] Chapple IL, Busby M, Clover H, Matthews R. Periodontal disease and systemic disease. J R Soc Med. 2014 Mar;107(3):94. doi: 10.1177/0141076813518770. No abstract available. PMID 24585887